CLINICAL TRIAL: NCT04768179
Title: A Randomized Clinical Trial to Investigate Safety & Efficacy of Low-dose Aspirin / Ivermectin Combination Therapy in Management of COVID-19 Patients
Brief Title: Safety & Efficacy of Low Dose Aspirin / Ivermectin Combination Therapy for Treatment of Covid-19 Patients
Acronym: IVCOM
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Makerere University (Other)
Collaborators: Ministry of Health, Uganda (Other Government); Mbarara University of Science and Technology (Other); Joint Clinical Research Center (Other)
Responsible Party: Principal Investigator, College of Health Sciences, Chair and Associate professor Department of Pharmacology and Therapeutics, Makerere University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IVCOM PROTOCOL VERSION 03
Record Dates: First submitted 2021-02-14; First posted 2021-02-24 (Actual); Last update posted 2021-02-24 (Actual); Status verified 2021-02

CONDITIONS: Covid19
Keywords: COVID-19 Therapies
MeSH Terms: conditions — COVID-19 | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Arm1 (Control group) (No Intervention): standard of care
- Arm 2 (Experimental): Drug: 3-dayIVM 200 mcg/kg/day/14-day 75mgASA/day + standard of care (intervention 1)
  Interventions: Drug: 3-dayIVM 200 mcg/kg/day/14-day 75mgASA/day + standard of care (intervention 1)
- Arm 3 (Experimental): 3-day Ivermectin 600 mcg/kg/day/14-day 75mgASA/day + standard of care (Intervention 2)
  Interventions: Drug: 3-dayIVM 200 mcg/kg/day/14-day 75mgASA/day + standard of care (intervention 1)

INTERVENTIONS:
Drug: 3-dayIVM 200 mcg/kg/day/14-day 75mgASA/day + standard of care (intervention 1) — Low dose aspirin for 14 days plus ivermectin at 200 mcg/kg/day or 600 mcg/kg/day for 3 days
  Other Names: 3-dayIVM 600 mcg/kg/day/14-day 75mgASA/day + standard of care (intervention 2)
  Arms: Arm 2; Arm 3

SUMMARY:
COVID-19, caused by the novel Severe Acute Respiratory Syndrome Corona Virus 2 (SARSCoV-2), has become a global pandemic. Fortunately, most of the COVID-19 cases confirmed are categorized as mild for whom home- based symptomatic management with monitoring of clinical deterioration is recommended. Despite providing symptomatic management, a therapeutic drug that would limit the course of infection is greatly needed to stop COVID-19 disease progression. Considering the current SARS-CoV-2 epidemiology and the legitimate rash towards appropriate therapies, our study seeks to evaluate the safety and efficacy of low dose aspirin and ivermectin combination therapy in COVID-19 patients.

DETAILED DESCRIPTION:
Micro clotting is to date reported as a major cause of death among COVID-19 patients. SARS-CoV-2 associated micro clotting results into acute respiratory distress syndrome (ARDS) and death. This micro-clotting cascade supports the potential role of anticoagulants like aspirin, heparin in the clinical management of COVID-19 patients. Other areas that could be considered for potential treatment of COVID-19 include drugs and analogues of drugs that have demonstrated potential in-vitro and or in-vivo activity against SARS-CoV-2 like hydroxychloroquine, azithromycin, lopinavir/ritonavir and remdesivir and ivermectin. Ivermectin has demonstrated broad-spectrum anti-viral activity and inhibition of the causative virus (SARS-CoV-2) with ability to cause a 5000-fold reduction in viral RNA within 48hrs.

Although aspirin and ivermectin do not exhibit any synergistic or potentiation at cellular level, a clinical additive effect resulting from combination therapy with low dose aspirin and ivermectin is plausible. There is no documented drug-drug interactions or other biological basis that contra-indicate co-administration of low dose aspirin and ivermectin.

We therefore propose, to explore the clinical use of combination anticoagulant: lower dose aspirin and the FDA-approved anti-parasitic drug: ivermectin, in treatment of COVID-19 patients in an exploratory randomized trial.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated informed consent form
* Willingness to comply with all study procedures and availability over the study duration *Patients aged above 18years to 64 years
* PCR positive for SARS-Cov-2 (COVID-19) from any of the MOH COVID-19 accredited testing laboratories
* Moderately ill COVID-19 patients score 3(Hospitalized with no oxygen therapy) to 4 (Hospitalized with oxygen by mask or nasal prongs) according to the WHO ordinal scale for clinical improvement which translates to moderate to severe COVID-19 patients according to the Ministry of Health Uganda COVID-19 disease category.

Exclusion criteria:

* Participants with known hypersensitivity to Ivermectin
* Clinical diagnosis of severe renal and hepatic impairment.
* Pregnancy or breast feeding.
* Co-treatment with either strong cytochrome p-450 inducers including: rifampicin, carbamazepine and barbiturates or inhibitors: isoniazid, clofazimine that might potentially affected ivermectin disposition and clinical outcomes
* Co-morbidities including asthma
* Loa loa as assessed by travel history to Angola, Cameroon, Chad, Central African Republic, Congo, DR Congo, Equatorial Guinea, Ethiopia, Gabon, Nigeria and Sudan in the last 4 years
* Persons clinically diagnosed with and receiving treatment for any diathesis and PUD
* Active participation in another clinical trial

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 490 (Estimated)
Dates: Start 2021-02-19 (Estimated); Primary Completion 2021-06-30 (Estimated); Study Completion 2021-09-30 (Estimated)

PRIMARY OUTCOMES:
SARS COV 2 Viral clearance | Day 14
  SARS COV 2 Viral load
World Health Organization COVID-19 ordinal improvement score | Day 14
  Minimum score is 0 (un infected, no clinical or virological evidence of infection) Maximum sore is 8 (death) Higher scores mean a worse outcome, low scores mean a better outcome

SECONDARY OUTCOMES:
Clinical recovery | Day 14
  disappearance or cessation of COVID-19 associated symptoms
Spectrum and severity of adverse events | Days one to day 14
  Adverse drug reactions
Maximum Plasma concentration | Days one to six
  average maximum ivermectin drug concentrations
Minimum Plasma concentration | Days one to six
  average minimum drug concentrations
Area Under the Curve | Days one to six
  Population drug concentrations from time of the first drug administration to the time when the last dose is eliminated

CONTACTS AND LOCATIONS:
Overall Officials: Jackson Mukonzo, PhD, Principal Investigator — Makerere University, college of Health Sciences

REFERENCES:
- [Derived] Fischer AL, Messer S, Riera R, Martimbianco ALC, Stegemann M, Estcourt LJ, Weibel S, Monsef I, Andreas M, Pacheco RL, Skoetz N. Antiplatelet agents for the treatment of adults with COVID-19. Cochrane Database Syst Rev. 2023 Jul 25;7(7):CD015078. doi: 10.1002/14651858.CD015078. PMID 37489818